CLINICAL TRIAL: NCT01555008
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Parallel Group Study to Evaluate the Pharmacodynamic and Pharmacokinetic Effects of LX4211 in Subjects With Type 2 Diabetes Mellitus and Moderate to Severe Renal Impairment
Brief Title: Study to Evaluate the Pharmacodynamic and Pharmacokinetic Effects of LX4211 in Subjects With Type 2 Diabetes and Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LX4211.1-107-DM; LX4211.107 (Other: Lexicon Pharmaceuticals, Inc.)
Record Dates: First submitted 2012-03-07; First posted 2012-03-15 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-09

CONDITIONS: Type 2 Diabetes Mellitus; Renal Impairment
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency | interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A (Experimental)
  Interventions: Drug: LX4211
- LX4211 Placebo (Placebo Comparator)
  Interventions: Drug: LX4211 Placebo

INTERVENTIONS:
Drug: LX4211 — Subjects will receive LX4211 once daily for 7 days
  Arms: Treatment A
Drug: LX4211 Placebo — Subjects will receive LX4211 placebo once daily for 7 days
  Arms: LX4211 Placebo

SUMMARY:
This Phase 1 study is intended to assess the pharmacodynamics (PD), pharmacokinetics (PK), safety and tolerability of LX4211 following once daily oral administration in subjects with type 2 diabetes mellitus (T2DM) and moderate to severe renal impairment.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 to ≤80 years of age
* History of T2DM for at least 6 months prior to screening
* Moderate to severe renal impairment and not actively on dialysis
* Willing and able to perform self-monitoring of blood glucose
* Willing and able to provide written informed consent

Exclusion Criteria:

* History of type 1 diabetes mellitus, diabetic ketoacidosis (within the previous 6 months), or diabetes resulting from pancreatic disorder or secondary diabetes (from acromegaly and/or Cushing's disease)
* Subjects who have received a renal allograft
* Subjects expecting to require dialysis or to undergo kidney transplantation within 3 months of study dosing
* Presence of active hepatic disease or clinically significant abnormal liver function tests at Screening or planned study Day -1
* Subjects with a history of heart attack, severe/unstable angina, or coronary revascularization procedure within 6 months prior to study Day -2
* History of clinically significant cardiac arrhythmias within 1 year prior to study Day -2
* Subjects with congestive heart failure
* Subjects with uncontrolled Stage III hypertension
* History of 2 or more emergency room visits, doctors' visits, or hospitalizations due to hypoglycemia within the 6 months prior to planned study Day -2
* History of alcohol or illicit drug abuse within 1 year prior to Screening
* History of human immunodeficiency virus (HIV), hepatitis B, or hepatitis C
* Major surgery within 6 months prior to planned study Day -2
* History of any malignancy within the last 5 years
* Triglycerides >1000 mg/dL at Screening or planned study Day -1
* History of any serious adverse reaction or hypersensitivity to an SGLT inhibitor
* Use of corticosteroids within 2 weeks prior to study Day 1
* Use of any investigational drug within 30 days prior to study Day 1, or investigational protein or antibodies within 60 days of Day 1
* Positive urine pregnancy test at Screening
* Positive urine screen for illicit drug abuse at Screening
* Prior exposure to LX4211

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2012-03; Primary Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in postprandial glucose | baseline to 7 days

SECONDARY OUTCOMES:
Number of subjects experiencing an adverse event | 7 days
Change from baseline in fasting plasma glucose | baseline to 7 days
Change from baseline in glucagon-like peptide 1 (Glp-1) | baseline to 7 days
Area Under Curve (AUC) | Days 1 and 7; predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, and 48 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Ike Ogbaa, M.D., Study Director — Lexicon Pharmaceuticals, Inc.
Locations (6):
- United States (6):
  - Lexicon Investigational Site, Anniston, Alabama
  - Lexicon Investigational Site, Chula Vista, California
  - Lexicon Investigational Site, Edgewater, Florida
  - Lexicon Investigational Site, Minneapolis, Minnesota
  - Lexicon Investigational Site, San Antonio, Texas
  - Lexicon Investigational Site, Renton, Washington

REFERENCES:
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818
- [Derived] Zambrowicz B, Lapuerta P, Strumph P, Banks P, Wilson A, Ogbaa I, Sands A, Powell D. LX4211 therapy reduces postprandial glucose levels in patients with type 2 diabetes mellitus and renal impairment despite low urinary glucose excretion. Clin Ther. 2015 Jan 1;37(1):71-82.e12. doi: 10.1016/j.clinthera.2014.10.026. Epub 2014 Dec 17. PMID 25529979